CLINICAL TRIAL: NCT01933282
Title: Phase II Study of MESA Chemotherapy in Patients With Natural Killer/T Cell Lymphoma
Brief Title: MESA Treatment for NK/T Cell Lymphoma
Acronym: MTN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Xie-qun Chen, Dean of Department of Hematology, Xijing Hosptial, Air Force Military Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MESA-NKT2013
Record Dates: First submitted 2013-08-16; First posted 2013-09-02 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Lymphoma, Extranodal NK-T-Cell
Keywords: MESA, chemotherapy,NK/T cell lymphoma
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MESA chemotherapy (Experimental): Methotrexate etoposide dexamethasone Polyehylene glycol-asparaginase Methotrexate 2g/ m2，IV d1 etoposide 100mg/ m2，VD d2，d3，d4 dexamethasone 20mg/ m2，VD d2，d3，d4，d5 Polyehylene glycol-asparaginase muscular injection 2500IU/ m2, d5
  Interventions: Drug: MESA chemotherapy; Drug: MESA

INTERVENTIONS:
Drug: MESA chemotherapy — Methotrexate 2g/ m2，IV d1 etoposide 100mg/ m2，VD d2，d3，d4， dexamethasone 20mg/ m2，VD d2，d3，d4, d5 Polyehylene glycol-asparaginase muscular injection 2500IU/ m2, d5
Drug: MESA — Methotrexate etoposide dexamethasone Polyehylene glycol-asparaginase

SUMMARY:
Study on the efficacy and safety of MESA chemotherapy for treating NK/T cell lymphoma

DETAILED DESCRIPTION:
Extranodal natural killer (NK)/T-cell lymphoma (ENKTL), nasal type, is a distinct and heterogeneous histopathologic subtype of non-Hodgkin lymphoma (NHL), accounting for 5%~10%. The frequency of ENKTL among NHL patients is significantly higher in Asia than in Western countries. Despite radiotherapy and chemotherapy, the prognosis for ENKTL patients is poor, with 5-year median survival time for primary nasal site was 5 years, for non-nasal extranodal sites 6 months. ENKTL is so aggressive and has high mortality rate and till now there is no standard therapy. In recent years SMILE chemotherapy has clinical efficacy and is one of first line therapy for ENKTL. However it is apparent that this regimen is extremely toxic with grade 4 neutropenia especially for Asian patients. On these grounds, new therapy MESA is used for Asian patients with ENKTL in order to achieve good efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis is NK/T cell lymphoma；
* At least one objective evaluation ( measurable ) lesions
* Age 15 ~ 60 years old, men and women are not limited
* ECOG(Eastern Cooperative Oncology Group）performance status 0~3，Expected to survive more than 3 months;
* Heart, kidney function in the normal range
* Liver function: transminase< 2 times the normal value
* pregnancy tests of women childbearing age must be negative; Men and women agree to use effective contraception during the treatment and the following year
* Before the test sign the written informed consent

Exclusion Criteria:

* The early use of methotrexate or/and L-asparaginase;
* Pregnant or nursing, psychiatric patients complicated with malignant tumor
* At the same time the application of other trial drug, drug contraindications exist in research;
* Serious infection or metabolic diseases
* Liver dysfunction, serum direct bilirubin, indirect bilirubin, transaminase 2 times higher than normal; serum total protein or albumin below normal;
* Renal insufficiency, creatinine clearance rate was 2 times higher than normal, especially the creatinine clearance rate is less than 30ml/min;
* Before entering the group, blood: White blood cell< 3×10E9/L; absolute neutrophil count<1.5×10E9/L; platelet<100×10E9/L ( bone marrow is not violated ); platelet count <75×10E9/L ( bone marrow invasion ); hemoglobin<100g/L.
* In the 6 months before entering the group, patients with uncontrolled or serious cardiovascular diseases, including myocardial infarction, III-IV class heart failure, uncontrolled angina or clinically significant pericardial disease, and diabetes and phlebitis;
* HIV antibody positive, HBsAg positive after antiviral HBV(hepatitis B virus) DNA titer in 104copies/ml the following groups. HIV antibody positive, HBsAg+ and DNA titer in 104copies/ml after antiviral HBV therapy
* Coagulation abnormalities.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
response criteria for CR(complete remission)by physical examination,lymph nodes masses and bone marrow test. | 24 week
  After 6 cycle of MESA treatment,response assessments for CR,PR(partial remission) and NR(no remission) should include appropriate imaging studies(CT,MRI and PET-CT) based on the type of study performed at initial workup, endoscopy with visual inspection, repeat biopsies and measurement of EBV DNA

SECONDARY OUTCOMES:
rate of survival | 1 year, 2 years, 3years
  prognosis assessment by rates of survival including PFS(Progression-Free-Survival) and OS(Overall survival)at 1 year,2 years,3 years after induction therapies and follow up therapies.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hemaology, Xi jing Hospital,The Fourth Military Medical University, Xi'an, Shaanxi, China